CLINICAL TRIAL: NCT02079623
Title: Implementation of Electroporation - NanoKnife as Treatment for Advanced Pancreatic Cancer.
Brief Title: Electroporation (NanoKnife) as Treatment for Advanced Pancreatic Cancer
Acronym: NanoKnife
Status: Completed | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Collaborators: Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Ole Thorlacius-Ussing, MD, DMSc, Professor of Surgery, MD, DMSc, Professor of Surgery, Aalborg University Hospital
Other Study IDs: PCaNanoK
Record Dates: First submitted 2014-03-04; First posted 2014-03-06 (Estimated); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic cancer; Electroporation; Nano knife treatment
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Electroporation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Pancreatic cancer: Patients with locally advanced pancreatic cancer.
  Interventions: Procedure: Electroporation/ Nano knife treatment; Device: NanoKnife

INTERVENTIONS:
Procedure: Electroporation/ Nano knife treatment
Device: NanoKnife

SUMMARY:
The aim for this study is to implement electroporation therapy (NanoKnife) treatment for patients with locally advanced pancreatic cancer. Electroporation therapy (NanoKnife) will be given in addition to standard chemotherapy.

DETAILED DESCRIPTION:
Pancreatic cancer has a very high mortality with a 5-year survival rate of less than 10 %. Even though pancreatic cancer accounts for only 2-3 % of all cancer cases, it is the 4th leading cause of cancer death. The best prognosis is observed in patients, where tumor is confined to pancreas, and where curative resection is feasible. This accounts for 5-12% of patients. After complete surgical resection, these patients have a median survival of 15-25 months and a 5-year survival rate of 8-15%. Approximately 40% of patients with pancreatic cancer have metastatic disease at time of diagnosis, a significantly worse prognosis with a median survival of 6-12 months and very low long-term survival (less than 1%). The remaining 40-50% of patients have locally advanced disease (LAPC) without metastases. It is not possible to do complete surgical resection of LAPC because the tumor is infiltrating the surrounding tissue or blood vessel. These patients also have a severe prognosis with a poor long-term survival and median survival time of approximately 12 months.

The majority of patients with LAPC are offered palliative chemotherapy as standard treatment. Few patients are offered downstaging with chemo-radiotherapy. In rare cases downstaging results in extensively tumor shrink which enables subsequently surgical resection. However, the majority of patients remain none-resectable and only candidates for palliative/symptomatic treatment.

Electroporation is a new local treatment of tumors. Tumor cells are exposed to series of direct current impulses with high voltage (1500 V / cm) of milliseconds duration. Electroporation was originally used to enhance the sensitivity of tumor cells to certain cytotoxic agents by increasing the permeability of the cell membrane. Later it was found that direct current at sufficiently high voltage can destroy the cell membrane of cancer cells without damaging surrounding connective tissue or blood vessels. By modulating the length of the impulses and voltage, this cell-killing effect is achieved without any significant heating of the tissue, which reduces the risk of thermal damage. Electroporation differs in this way from other forms of local treatment such as radiofrequency ablation (RFA), which acts through the heating and coagulation of tissue.

The aim for this study is to implement electroporation therapy (NanoKnife) treatment for patients with locally advanced pancreatic cancer. Electroporation therapy (NanoKnife) will be given in addition to standard chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients above 18 years old, who have given informed consent to treatment with electroporation
2. Performance status <= 2 and meets one of the items below
3. Patients diagnosed with LAPC, who are not candidate to primary curative surgical treatment due to tumor invasion in surrounding blood vessels or adjacent organs
4. Patients, who have received oncological treatment with the aim of downstaging and the tumor still is deemed none-resectable

Exclusion Criteria:

1. Patients with pacemaker or similar electrostimulator (TNS, anal sphincter stimulators ect.)
2. Patients for whom the anesthesia involves high risk (ASA- IV)
3. Estimated survival of less than 3 months
4. Metallic stent in the biliary tract, which can not be removed or changed to plastic stent.
5. Performance status > 2.
6. Pregnancy
7. Epilepsy or other condition involving convulsions
8. Inability to give informed consent.
9. Patients with inability to cooperate for treatment and follow-up
10. Severe heart disease
11. Patients with a tumor larger than 5 cm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with locally advanced pancreatic cancer
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Tumor response | 24 months follow-up
  According to RECIST criteria (PET-CT)

SECONDARY OUTCOMES:
CA-19-9 | 24 months follow up
  CA-19-9 measurement every 3 months
Overall survival | 24 months follow-up

OTHER OUTCOMES:
Pain registration | 24 months follow up
  Pain registration pre- and post NanoKnife treatment using the visual analogue scale of 0 to 10. Higher numbers refer to worse pain.

CONTACTS AND LOCATIONS:
Overall Officials: Ole Thorlacius-Ussing, Prof., cons., dr. med, Study Chair — Department of Gastroinstestinal Surgery, Aalborg University Hospital
Locations (1):
- Surgical Department of Gastroenterology, Aalborg University Hospital, Aalborg, Nothern Jutland, Denmark